CLINICAL TRIAL: NCT06535919
Title: Substance Use Treatment and Its Role in Supporting Social Cognition
Acronym: SUE
Status: Recruiting | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Madison Roopchand, Psychology Trainee, MS, Nova Southeastern University
Other Study IDs: 2024-286
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Substance Use; Empathy
Keywords: substance use, empathy
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RUP: Individuals receiving TAU from RUP
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Treatment as Usual — Individuals will receive residential level of care followed by treatment at their partial hospitalization program.

SUMMARY:
This study aims to assess changes in empathy levels before and after residential treatment among individuals with substance use disorders.

DETAILED DESCRIPTION:
Despite the lack of a consensus on the conceptualization of empathy among researchers and practitioners, psychologists generally agree that empathy and valuable interpersonal relations are contingent upon the willingness to understand another's perspective as well as share feelings and experiences. Adults with a variety of substance use disorders (SUDs) experience impairments in various facets of empathetic processing compared to healthy controls. Impairments in empathy could lead to a weak therapeutic alliance, lower adherence to treatment, and higher relapse rate. Furthermore, the therapeutic relationship has been described as one of the strongest predictors of treatment drop-out for patients with SUDs. In addition, an impaired ability to relate to and understand the affective and mental state of others may contribute to key typologies of patients with SUDs including, impulsivity, aggression, and antisocial behavior. Review of literature emphasizes a need for research into an understudied, yet modifiable factor of empathy in the trajectory of SUDs. Particularly, identifying specific psychotherapeutic techniques capable of improving the expression of empathy in these patients. Given the importance of empathetic ability in optimal social functioning, understanding whether empathetic impairments improve with treatment is important to achieve the best treatment outcomes for individuals struggling with SUDs.This study will help improve the knowledge and understanding of how substance use treatment affects empathy, as measured by gains in empathetic ability in treatment seeking individuals. To date, there are no reported studies that examined the impact of residential SU treatment on empathy. The study will be an observational quasi-experimental design that utilizes a pre-test and post-test to examine change in empathy for recently detoxed substance use patients and a follow-up assessment to monitor long term outcomes. The results of this study will further our understanding of treatment's potential role in cultivating a fundamental interpersonal skill, empathy.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for a substance Use Disorder, receiving treatment at Recovery Unplugged Addiction Treatment Center, at least 18 years of age.

Exclusion Criteria:

* Neurological disorder, severe cognitive impairment, comorbid thought disorder such as schizophrenia, failure to complete detox period,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual receiving treatment at a local addiction treatment center.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-10-22 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
empathy | pre to post treatment and 2 month post treatment follow-up (4 months total)
  The Empathy Quotient-Short (EQ-Short) is a self-report questionnaire designed to assess individual differences in empathy. It is used to measure levels of empathy, including affective, cognitive, and total empathy. The unit of measure for the outcome is the total empathy score derived from responses to 22 items, with each item rated on a 4-point Likert scale ranging from 1 ("I strongly disagree") to 4 ("I strongly agree"). For example, one of the items asks, "I can pick up quickly if someone says one thing but means another." This scale is designed to assess various facets of empathy, including the ability to recognize emotions in others (cognitive empathy) and the ability to share or respond to those emotions (affective empathy). Previous multivariate analyses suggest that the Empathy Quotient-Short is a reliable and adequate tool for assessing individual differences in empathizing.

SECONDARY OUTCOMES:
differences in empathy gains by sex | pre and post treatment, 2 month post treatment follow-up (4 months total)
  A secondary outcome of this study is to assess differences in empathy gains between men and women. Specifically, the study will examine how levels of empathy change over time as a function of sex. Empathy will be measured using the Empathy Quotient-Short (EQ-Short), which evaluates affective, cognitive, and total empathy. The unit of measure for this outcome is the change in total empathy scores before and after the intervention, with the empathy score calculated based on participants' responses to 22 items on a 4-point Likert scale. The analysis will focus on comparing the magnitude of empathy changes between male and female participants to identify potential differences in the extent to which empathy increases for each sex. This will provide insight into whether the intervention leads to varying levels of empathy development based on sex.

OTHER OUTCOMES:
Substance Use | Baseline and 2 months post treatment follow-up
  The Brief Addiction Monitor (BAM) (Cacciola et al., 2013) is a 17-item self-report questionnaire used to assess substance use behaviors. The tool includes three subscales: (1) Current Use, (2) Current Risk, and (3) Protective Factors. The unit of measure for this outcome is the frequency and intensity of substance use behaviors, as assessed by responses to individual items within the subscales. Of the 17 items, 16 are single-response, and one is a multi-response item regarding drug use frequency. Specifically, ten items are rated on a 5-point Likert scale (0 to 10), denoting the number of days participants engaged in substance-related behaviors. Five items are rated on a 5-point ordinal scale ranging from (1) "Not at All" to (5) "Extremely," one item uses a binary scale (Yes/No), and one item is rated from "poor" to "excellent." At Time 2 and Time 3 assessments during treatment, the substance use-related items will be omitted.
Social Support | Baseline and post treatment as well as 2 month post treatment follow-up
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item self-report questionnaire used to assess an individual's perception of social support from three key sources: family, friends, and a significant other. The unit of measure for this outcome is the perceived level of social support, with responses rated on a 7-point Likert scale ranging from (1) "I very strongly disagree" to (7) "I very strongly agree." For example, one item asks, "There is a special person who is around when I am in need." The Multidimensional Scale of Perceived Social Support has demonstrated strong internal consistency, test-retest reliability, validity, and a stable factorial structure across multiple studies, making it a reliable tool for measuring perceived social support.
Therapeutic Alliance | Baseline, pre-discharge from residential and at PHP treatment pre-discharge
  The Working Alliance Inventory-Short Form (WAI-SF) is a 12-item self-report questionnaire used to assess the working alliance in therapy. The measure will be completed by both participants and therapists to evaluate their perceptions of the working relationship. The unit of measure for this outcome is the perceived strength of the working alliance, with responses rated on a 5-point Likert scale ranging from (1) "never" to (5) "always." For example, one item asks, "My therapist and I are working towards mutually agreed upon goals." The Working Alliance Inventory-Short Form consists of three subscales: (1) Goals (agreement on therapy goals), (2) Tasks (agreement on therapy tasks), and (3) Bond (the emotional connection between therapist and client). The WAI has demonstrated strong psychometric properties, including high internal consistency and good construct validity, making it a reliable tool for measuring the quality of the therapeutic alliance.
Report of therapist Emapthy | Baseline, pre-discharge from residential , pre-discharge from PHP
  The Barrett-Lennard Relationship Inventory-Empathy (BLRI-Empathy) is a self-report measure of empathy that is widely used in therapeutic settings. The unit of measure for this outcome is the perceived level of empathy, with participants rating their perception of the therapist's empathy and therapists rating their perception of the patient's empathy. The empathy subscale consists of 16 items (e.g., "My therapist understands me"), which are rated on a 6-point Likert scale ranging from (-3) "I strongly feel that it is not true" to (3) "I strongly feel that it is true." The Barrett-Lennard Relationship Inventory-Empathy has demonstrated strong internal consistency, test-retest reliability, and both convergent and divergent validity, as well as predictive validity in past research, supporting its use as a reliable tool for assessing empathy in therapeutic relationships.
Reflective Functioning | Baseline, Pre-discharge residential, pre-discharge PHP, two month follow-up
  The Reflective Functioning Questionnaire (RFQ) is a self-report questionnaire designed to assess an individual's capacity for mentalization-the ability to understand and interpret one's own and others' behaviors based on underlying mental states. The unit of measure for this outcome is the level of reflective functioning, with higher scores indicating greater mentalization capacity. The questionnaire consists of 8 items (e.g., "Sometimes I do things without really knowing why"), which are rated on a 7-point Likert scale from (1) "I strongly agree" to (7) "I strongly disagree." Higher total scores reflect higher reflective functioning. The Reflective Functioning Questionnaire has demonstrated good reliability and test-retest consistency, making it a valid and reliable tool for measuring reflective functioning.
Therapeutic Orientation Processes | Baseline, pre-discharge from residential, pre-discharge from PHP
  The Therapy Process Observational Coding System (TPOCS) is a coding system designed to assess the therapeutic process in psychodynamic and cognitive behavioral therapies. The unit of measure for this outcome is the relative difference in therapeutic processes between psychodynamic and cognitive behavioral therapies, with higher scores indicating a greater emphasis on psychodynamic interventions. The measure consists of 22 items that capture therapist interventions and processes unique to each therapy type. For example, an item might read, "My therapist emphasizes my feelings to help me experience them more deeply." Responses are rated on a 7-point Likert scale ranging from (1) "not at all" to (7) "very much so." The TPOCS will be analyzed using the relative psychodynamic therapies difference score (psychodynamic therapies minus cognitive behavioral therapies), which accounts for various sources of measurement error.
Confidence to Participate | Baseline, pre-discharge from residential and at PHP treatment pre-discharge
  To assess a participant's confidence and likelihood of participating in the upcoming assessment, we use a single-item measure: "On a scale from 1 to 10, how confident are you in your ability to participate in the upcoming assessment, with 1 being 'Not confident at all' and 10 being 'Extremely confident'?" This question will help to gauge the participant's self-reported readiness and assurance about engaging in the assessment process, providing a straightforward indicator of their anticipated involvement and commitment.
Participation in Additional Services | Two month follow-up post treatment
  To assess a participant's participation in professional treatment or self-help involvement two items will be used: "Since the conclusion of your treatment at the partial hospitalization program, how frequently have you engaged in any self-help activities?" and "Since the conclusion of your treatment at the partial hospitalization program at recovery unplugged, how frequently have you engaged in any other professional treatment?" The items are measured on a 5-point Likert scale denoting the number of days engaged in additional services over the past 60 days. This assessment will help gauge the participant's self-reported engagement in additional services, providing a straightforward indicator of their involvement post-intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Recovery Unplugged, Fort Lauderdale, Florida
  - Recovery Unplugged, Lake Worth, Florida

IPD SHARING:
Plan to Share IPD: Undecided